CLINICAL TRIAL: NCT06035107
Title: Clinical Validation of Contactless Radar Blood Pressure Device
Brief Title: Contactless Radar Blood Pressure Validation
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 160695; IRAS ID: 328944 (Other: HRA)
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 25 participants will undergo radar blood pressure tests during an MRI scan of the heart. In these participants, a point of care blood test will be taken to assess kidney function using the StatSensor Xpress Creatinine monitor (Nova Biomedical, USA). Additional blood tests will also be collected for storage and future DNA and small molecule analysis.
  The other participants will not have biospecimens stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Comparing radar and auscultatory blood pressure: 25 participants will be recruited from a specialist hypertension clinic. These participants will undergo the following tests:
  1. Questionnaire: The participant will be asked to complete a clinico-demographic questionnaire. This includes their demographic data and past medical history.
  2. Measurement of height, weight and heart rate
  3. Measurement of blood pressure using the radar device and using a cuff (called manual auscultation)
  4. End of visit.
  Interventions: Diagnostic Test: Radar blood pressure device
- Comparing radar and invasive blood pressure: Participants will be recruited from a list of patients scheduled to attend the Royal Free Hospital catheterisation laboratory for a clinically-indicated invasive angiogram that was booked by their consultant. 50 participants aged 18 and over will be recruited.
  The radar blood pressure measurements taken during the angiogram will not impact on the procedure or standard clinical care which the participant will receive. The duration of the visit is determined by the duration of the coronary angiogram and that is decided by the clinical care team. Participants will have the following tests:
  1. Collection of baseline data including past medical history, current medication, height, weight and baseline ECG
  2. Measurement of invasive blood pressure and radar blood pressure simultaneously before the rest of the procedure
  3. End of visit.
  Interventions: Diagnostic Test: Radar blood pressure device
- Testing if the radar device can measure blood pressure in the MRI scanner: First we will develop a radar blood pressure device that can be used in the MRI scanner.
  When this device has been proven to be safe, we will recruit 25 participants to have the following tests:
  1. A questionnaire. The participant will be asked to complete a clinic-demographic questionnaire including their demographic data and past medical history.
  2. Collection of blood test to assess kidney function. Additional blood tests will also be collected for storage and future analysis.
  3. A cardiac MRI scan. Blood pressure will be measured at 5 minute intervals during the scan using an oscillometric cuff around the right upper arm. The radar device will measure blood pressure in a contactless way at the same time.
  4. End of visit.
  Interventions: Diagnostic Test: Radar blood pressure device
- Testing if the radar device can measure blood pressure during exercise: We will recruit 50 participants the have the following tests:
  1. Questionnaire: The participant will be asked to complete a clinico-demographic questionnaire. This includes their demographic data and past medical history.
  2. Measurement of heart rate, breathing rate and oxygen saturations.
  3. Recording a heart tracing called an ECG
  4. Participants will then perform 5-10 minutes of exercise, either repeated sit-to-stand movements or using a bike ergometer. Blood pressure will be measured using a cuff and the radar device at regular intervals
  5. Participants will then have a heart scan called an echocardiogram during which time the radar blood measurements will also be collected.
  6. End of visit.
  Interventions: Diagnostic Test: Radar blood pressure device

INTERVENTIONS:
Diagnostic Test: Radar blood pressure device — The radar blood pressure device will be compared with other traditional blood pressure measurement methods.

SUMMARY:
The goal of this observational study is to learn how accurately blood pressure can be measured using a contactless radar device.

The main questions the study aims to answer are:

1. how does blood pressure measured using radar compare with blood pressure using a cuff in patients with known high blood pressure?
2. how does blood pressure measured using radar compare with invasive blood pressure during a coronary angiogram?
3. can the radar blood pressure machine be used to measure blood pressuring during an MRI scan of the heart?
4. can the radar blood pressure machine be used to measure blood pressure during exercise?

Participants in this study will have the following tests:

Group 1: blood pressure measured with the radar device and a cuff when resting Group 2: blood pressure measured with the radar device and by placing a small tube inside the arteries of the wrist (during a clinical procedure) Group 3: blood pressure measured with the radar device and a cuff during a cardiac MRI scan Group 4: blood pressure measured with the radar device and a cuff during exercise

DETAILED DESCRIPTION:
High blood pressure is the biggest risk factor for heart attacks and strokes. There are several machines available for measuring blood pressure, but most of them need to contact the skin causing discomfort from the inflatable cuff or risking the transmission of infections from reusing cuffs. There are also situations where the cuff machines are inaccurate, such as in older people or during exercise. Therefore, the investigators are trying to develop an accurate contactless system for measuring blood pressure.

The investigators have used advanced but safe radar to create a small machine with a camera that can measure blood pressure from a distance without the need to contact the participant's skin anywhere. It works by detecting tiny movements and changes on the skin produced from the heartbeat and pulse that cannot be seen with the human eye. The investigators want to study how accurate our radar blood pressure machine is by comparing it to other traditional methods of measuring blood pressure.

Firstly, radar blood pressure will be compared to auscultatory blood pressure (a blood pressure system using a cuff) in a group of 25 participants at rest attending a specialist blood pressure clinic. This is currently the internationally recommended method for validating new blood pressure devices.

Then radar blood pressure will be compared with invasive blood pressure (measured inside the arteries by a small tube) in 50 participants undergoing clinically-indicated cardiac catheterisation at the Royal Free Hospital.

Next a radar device capable of measuring blood pressure in participants lying inside the cardiovascular magnetic resonance (CMR) scanner will be developed. The radar blood pressure derived in the CMR scanner will be compared to oscillometric blood pressure in 25 participants (a cuff-based BP system that is currently used in patients being scanned). Finally, radar-BP will be compared with oscillometric BP in 50 participants during exercise including sit-to-stand movements and using a bike ergometer.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Age > 18 years old
* under the care of the complex hypertension clinic
* able to take auscultatory blood pressure from right arm

Group 2:

* Age >18
* has been selected to undergo invasive coronary angiogram by a consultant cardiologist

Group 3:

* Age >18
* willing to undergo a cardiac MRI scan

Group 4:

- Age > 18

Exclusion Criteria:

Group 1

* anyone unable to consent
* inaudible Korotkoff K1/K5 sounds
* systolic BP difference >12 mmHg and/or diastolic >8 mmHg in any of the auscultatory measurements during the validation study
* contraindication to cuff-based BP measurement e.g. lymph node clearance on right side

Group 2:

* anyone unable to consent
* anyone in whom right radial arterial access cannot be obtained (e.g. severe skin abnormality such as scleroderma)
* known arterio-venous malformation or fistulas in right arm
* any contraindication to an invasive angiogram such as severe frailty

Group 3:

* anyone unable to consent
* anyone with a classical contraindication to an MRI study such as known metal fragments allergy to used contrast
* high degree heart block
* asthma

Group 4:

* anyone unable to consent
* anyone with exertional chest pain or known uncontrolled angina
* anyone with a known positive cardiac stress test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: participants under the specialist hypertension clinic at the Royal Free Hospital Group 2: participants who have been selected to undergo an angiogram by a consultant cardiologist Group 3 and 4: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Radar blood pressure compared with blood pressure measured by manual auscultation | 3 years
  To determine if the radar module can derive accurate blood pressure measurements when compared against non-invasive blood pressure measurements by manual auscultation in a group of participants with known hypertension.

SECONDARY OUTCOMES:
Radar blood pressure compared with blood pressure measured invasively | 3 years
  To compare the blood pressure measurements from the radar BP device with invasive blood pressure measurements obtained at the time of coronary angiography

OTHER OUTCOMES:
Radar blood pressure compared with oscillometric blood pressure during a cardiac MRI scan | 3 years
  To compare the radar BP measurements with readings from an oscillometric cuff during a cardiac MR scan
Radar blood pressure compared with oscillometric blood pressure during exercise | 3 years
  To compare the radar BP measurements with readings from an oscillometric cuff during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Captur, PhD, Principal Investigator — University College, London
Locations (1):
- UCL Bloomsbury Centre for Clinical Phenotyping, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No